CLINICAL TRIAL: NCT02120755
Title: A Randomized Comparison of AmnioClear™ Human Allograft Amniotic Membrane vs. Moist Wound Dressing in the Treatment of Diabetic Wounds
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Never Started
Sponsor: Liventa Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Amn-DFU-01
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Foot Ulcers; Wound Care
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AmnioClear™ (Active Comparator): AmnioClear™ Human Allograft Amniotic Membrane
  Interventions: Biological: AmnioClear™ Human Allograft Amniotic Membrane
- Standard of Care (No Intervention): Standard moist wound dressing (saline wet-to-moist or a hydrogel dressing)

INTERVENTIONS:
Biological: AmnioClear™ Human Allograft Amniotic Membrane
  Arms: AmnioClear™

SUMMARY:
This research project is testing a product called AmnioClear™ which is an amniotic membrane graft processed for Liventa Bioscience formerly AFCell Medical. AmnioClear™ allograft human amniotic membrane is regulated solely under section 361 of the Public Health Service Act.

The purpose of the study is to see if this treatment works to accelerate the healing time of chronic wounds.

ELIGIBILITY:
Inclusion Criteria:

* Stable Type I or II diabetes mellitus
* At least one chronic diabetic ulcer
* Full-thickness ulcer size from 1-8 cm2.

Exclusion Criteria:

* Concurrent use of corticosteroids, NSAIDs immuno-suppressive or cytotoxic agents
* Bleeding disorders
* Ulcer with muscle, tendon, capsule or bone involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Reduction in Wound Size | 12 Weeks
  Clinical assessment of wound healing in terms of the reduction in size and shape of the wound over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States